CLINICAL TRIAL: NCT06267755
Title: Efficacy of Extracorporeal Shockwave Therapy on Ultrasonography Changes of Upper Trapezius Myofascial Trigger Points in Patients With Non Specific Neck Pain
Acronym: MTP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004884
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain
Keywords: Extracorporeal Shockwave Therapy; Ultrasonography Changes; Non Specific Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: extracorporeal shockwave and traditional therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Shockwave therapy (Experimental): Thirty patients will receive Extracorporeal Shockwave therapy and Traditional physical therapy three times per week for six consecutive weeks.
  Interventions: Other: Extracorporeal Shockwave therapy; Other: Traditional physical therapy
- Traditional physical therapy (Active Comparator): Thirty patients will receive Traditional physical therapy three times per week for six consecutive weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Extracorporeal Shockwave therapy — the patients will receive Extracorporeal Shockwave therapy sessions by 600 impulses with 1.6 bar pressure at a frequency of 8 Hz on site of the upper trapezius
  Arms: Extracorporeal Shockwave therapy
Other: Traditional physical therapy — the patients will receive Traditional physical therapy in the form of Integrated neuro-muscular inhibition technique + posture correction and scapular stabilization exercises.

SUMMARY:
this study will be conducted to investigate the effect of Extracorporeal Shockwave Therapy on Ultrasonography Changes of Upper Trapezius Myofascial Trigger Points in Patients With Non Specific Neck Pain

DETAILED DESCRIPTION:
Neck pain is one of the most commonly reported musculoskeletal disorders. The prevalence for neck pain varies between 16.7% and 75.1% in the general population. Up to 67% of world's population may present chronic non-specific neck pain at least once in their lives. The upper trapezius is probably the muscle most often beset by trigger points, it is indicated that the upper trapezius is the most sensitive of 8 different muscles (upper trapezius, pectoralis major, levator scapulae, teres major, supraspinatus, gluteus medius, infraspinatus, paraspinal) to the pressure of an algometer.Recently, the extracorporeal shock wave has been widely known to be an effective therapeutic modality in myofascial pain syndrome treatment and a systematic review provided promising insight into the effectiveness of ESWT in Myofascial pain syndrome treatment. sixty patients with non specific neck pain will be assigned randomly to two groups; first one will receive shock wave therapy and traditional therapy and the second one will receive traditional therapy only for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients receiving a diagnosis of non-specific neck pain with upper trapezius myofascial trigger points by an orthopaedist physician.
* Body mass index of participants was normal less than (30 kg/m2)(Al-asadi, 2018).
* Age over 18 years.
* Presence of taught band.
* Presence of hyper irritable spot in a taught band, and reproduction of the typical referred pain pattern of the myofascial trigger point in response to compression

Exclusion Criteria:

* Having signs and symptoms of neurological disorders that cause nerve root compression.
* Headache as a consequence of specific headache diagnosis.
* Having a history of specific signs of malignancy, or infection.
* Having a history of trauma with or without proven structural disorders in the region of the neck, shoulder, and head (e.g. whiplash).
* Having signs and symptoms of cerebrovascular insufficiency.
* Having a severe chronic disease of the locomotor system (e.g. polyarthritis, muscular disease
* Any participant with contraindications to shock wave therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
muscle thickness | up to six weeks
  Ultrasonography device will be used to assess muscle thickness
hypoechoic area intensity | up to six weeks
  An ultrasonography device will be used to assess the hypoechoic area intensity

SECONDARY OUTCOMES:
neck disability | up to six weeks
  Arabic version of neck disability index will be used to measure neck disability. It consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. 5 Each item is scored from 0 (no disability) to 5 (total disability). The maximum possible score is 50.
pressure pain threshold | up to six weeks
  Digital algometer will be used to measure pressure pain threshold
cervical range of motion | up to six weeks
  The cervical range of motion (CROM) device will be used to measure cervical ROM
pain intensity | up to six weeks
  The visual analog scale (VAS) will be used to measure pain intensity. it is a10 cm line, oriented vertically or horizontally, with one end representing "no pain" and the other end representing pain as bad as it can be